CLINICAL TRIAL: NCT07358286
Title: THE EFFECT OF KOLCABA'S COMFORT THEORY-BASED MOBILE EDUCATION ON COMFORT LEVELS OF OSTOMY PATIENTS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: MOBILE EDUCATION AND COMFORT IN OSTOMY PATIENTS
Acronym: STOMA-PLUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gökçe Nur Taşkıran, PhD Student, Nursing, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EGEU_PHD_STOMA_2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Stoma; Ostomy; Mobile Application
Keywords: Ostomy Care; Mobile Health; Kolcaba's Comfort Theory; Nursing

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, controlled, parallel-group, single-blind intervention study. Participants will be randomly assigned to either an intervention group receiving comfort theory-based mobile education or a control group receiving standard care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Participants are not informed about their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive standard postoperative care only, without the mobile education intervention.
- Experimental Group (Experimental): Participants in the experimental group will receive a mobile education program based on Kolcaba's Comfort Theory, including animation-based stoma care education, in addition to standard postoperative care.
  Interventions: Behavioral: Mobile Education Program Based on Kolcaba's Comfort Theory

INTERVENTIONS:
Behavioral: Mobile Education Program Based on Kolcaba's Comfort Theory — The intervention consists of a mobile education program based on Kolcaba's Comfort Theory. The program includes animation-based educational content on stoma care, pouch changing, peristomal skin care, and postoperative self-care. The mobile education is designed to support patients in managing their stoma and to improve their overall comfort levels.
  Other Names: The intervention consists of a mobile education program based on Kolcaba's Comfort Theory, including animation-based stoma care education. The program provides information on stoma care, pouch changin
  Arms: Experimental Group

SUMMARY:
Purpose of the Study

This study aims to understand whether a mobile education program can improve comfort levels in people living with a stoma. A stoma is a surgical opening created on the abdomen to allow stool or urine to leave the body. Living with a stoma can affect daily life in many ways, including physical comfort, emotional well-being, social life, and the home environment.

The education program used in this study is based on Kolcaba's Comfort Theory. This theory focuses on comfort as a whole and includes physical, emotional, social, and environmental aspects of a person's life. The study will compare people who receive mobile education with those who receive standard hospital care only.

Who Can Take Part

Adults aged 18 years and older who are scheduled to have colostomy, ileostomy, or urostomy surgery may take part in this study. Participants must be able to communicate in Turkish, read and understand written information, and agree to join the study voluntarily.

People with severe cognitive problems, serious communication difficulties, or major vision or hearing problems will not be included.

What Will Happen in the Study

Participants will be randomly assigned to one of two groups:

Mobile Education Group

Standard Care Group

Both groups will receive routine care provided by the hospital.

Participants in the mobile education group will also receive access to a mobile application designed specifically for people with a stoma. This application includes:

Easy-to-understand information about stoma care

Animated educational videos showing step-by-step stoma care practices

Guidance on skin care, pouch changing, and hygiene

Information on common problems and when to seek medical help

Reminders to support daily stoma care routines

The mobile application can be used on smartphones and does not include diagnosis or treatment. It is for education and support only.

Participants in the standard care group will receive usual hospital education and care. After the study is completed, they will also be offered the mobile education program.

What Participants Will Be Asked to Do

All participants will be asked to answer questionnaires that measure comfort levels at several time points:

Before surgery

One day after surgery

Fifteen days after discharge (by phone)

One month after surgery (during a clinic visit)

Participants in the mobile education group will be shown how to use the application and may use it as often as they wish. Researchers may contact participants to ask about their experience using the app and to identify any difficulties.

Possible Benefits

Participants may gain better understanding of stoma care and feel more confident managing daily life with a stoma. The mobile education program may help reduce discomfort, support emotional well-being, and improve overall quality of life.

The results of this study may help healthcare professionals develop better education tools and support programs for people living with a stoma.

Risks and Safety

This study does not involve experimental medical treatments. The mobile application provides education only. Personal data will not be collected through the app, and all information will be kept confidential. Participants may leave the study at any time without affecting their medical care.

Why This Study Is Important

Access to stoma care education can be limited due to time constraints, staff availability, and hospital resources. Mobile education may provide an easy and accessible way for people to receive reliable information whenever they need it.

This study will help determine whether a comfort-focused mobile education program can support people living with a stoma and improve their overall comfort and well-being.

DETAILED DESCRIPTION:
Stoma creation is one of the most commonly used surgical interventions in cancers of the urinary or gastrointestinal system, inflammatory bowel diseases, and traumatic conditions (United Ostomy Associations of America, 2021). The most common indications for stoma formation include Crohn's disease, diverticulitis, colon and rectal cancers, bladder cancer, adenomatous polyposis, neurogenic bladder dysfunction, ulcerative colitis, and traumatic ileus. The primary purposes of stoma creation are to prolong life expectancy, eliminate pathological conditions, and improve quality of life (Aksoy & Çavdar, 2015; Ayalon & Bachner, 2019; Barnwell, 2015; Burch, 2015; Tonolini, 2019; Wound, 2018).

Depending on the indication, a stoma may be temporary or permanent (Aksoy & Çavdar, 2015; Ayalon & Bachner, 2019). Temporary stomas account for approximately forty percent of all stomas. Colorectal cancers are the most common reason for permanent stoma creation. This type of cancer is among the five most common cancers in Türkiye (Ayalon & Bachner, 2019). According to the 2024 data from the World Health Organization's International Agency for Research on Cancer, colon cancer ranks second among cancer-related causes of death worldwide (World Health Organization, 2024).

It is estimated that approximately two million people worldwide live with a stoma, with around seven hundred thousand residing in Europe (Claessens et al., 2015). In the United States, an average of one hundred thirty thousand people undergo ostomy surgery each year, and it is estimated that approximately one million individuals live with urinary or fecal diversions (United Ostomy Associations of America, 2021). The number of individuals living with an ostomy is reported to exceed one hundred thousand in the United Kingdom and range between seven hundred twenty-five thousand and one million in North America (İncesu & Ulupınar, 2022). In Türkiye, the exact number of individuals living with a stoma is not clearly known (Çevik et al., 2020). However, due to the high prevalence of colorectal cancers, the rate of stoma creation is estimated to be considerable (Ayık et al., 2023).

After stoma surgery, individuals may experience both positive and negative physical, social, and psychological effects (Ayaz et al., 2008; Pinquart, 2010; Grant et al., 2013; Alptekin et al., 2023). Although survival rates increase significantly following stoma surgery, many complications may also occur. These complications can reduce quality of life, negatively affect physical and mental health, increase hospital length of stay, raise morbidity rates, and lead to higher healthcare costs. Such complications represent some of the negative consequences of living with a stoma (Kuzu et al., 2002; Karadağ et al., 2011; Salvadalena, 2013; Goldberg et al., 2018; Tonolini, 2019; Ayık et al., 2020; Hsu et al., 2020).

Adapting to life after stoma surgery is a challenging and time-consuming process. During this period, individuals need accurate education and adequate social support. Studies have shown that individuals who receive sufficient and appropriate education on stoma care demonstrate higher levels of adaptation compared to those who do not (Aminisani et al., 2017). Nurses play a crucial role in the adaptation process during both preoperative and postoperative periods. Their responsibilities include providing education, offering counseling services, informing individuals with a stoma, building self-confidence, and supporting post-discharge care (Duluklu & Çelik, 2019).

The role of stoma and wound care nurses in stoma management is invaluable. However, not all hospitals in Türkiye employ stoma and wound care nurses, and even in institutions where they are available, providing continuous care across all shifts is often not possible (Ayık et al., 2023). Kang et al. (2025) reported that individuals with a stoma face complex physiological, psychological, and social challenges during the postoperative period. The same study emphasized that holistic care and continuous support from healthcare professionals play a critical role in adaptation to life with a stoma.

Adaptation to stoma is influenced by factors such as individual competencies, demographic characteristics, and social support systems (Öztürk, 2019; Akil & Taylan, 2020). Similar to findings in other countries, studies conducted in Türkiye indicate that quality of life is negatively affected after stoma creation (Duluklu et al., 2019). Individuals living with a stoma frequently experience issues such as odor, leakage, body image disturbance, constipation, diarrhea, difficulty bathing, challenges related to sexuality, travel, and religious practices, all of which negatively affect quality of life (Duluklu et al., 2019).

Several international studies have reported reduced quality of life among individuals living with a stoma. In Brazil, Salomé et al. (2019) reported a mean quality of life score of 26.16 out of 105. In Malaysia, Thamilselvam et al. (2020) found that many participants reported family neglect, lack of sexual intimacy, limited social participation, and feelings of social exclusion. In the Netherlands, Gooszen et al. (2021) reported that twelve percent of individuals isolated themselves within the first three months after surgery, while seventy-two percent experienced problems related to clothing, diet, skin irritation, and leakage. Similarly, studies conducted in Iran and other countries have highlighted challenges related to nutrition, psychological changes, social relationships, physical activity, religious practices, and economic difficulties (Dabirian et al., 2022; Brady et al., 2025).

One of the key factors influencing quality of life among individuals living with a stoma is comfort. Comfort is considered a fundamental human need and a desired state throughout life (Yücel, 2011; Orkun et al., 2017). In nursing, comfort involves identifying patient needs, implementing appropriate interventions, and evaluating outcomes. Comfort is a complex, holistic, and individualized concept closely associated with the art of nursing (Çınar Yücel, 2011). Nursing care that prioritizes comfort in the postoperative period may accelerate recovery and improve overall well-being (Akalın et al., 2020).

Advancements in technology have increasingly contributed to disease management and quality of life assessment in healthcare. Mobile health applications installed on smartphones provide practical tools for disease management, follow-up, and patient support. These technologies facilitate home-based monitoring, reduce hospital workload, and lower healthcare costs (Langer et al., 2021). Studies have shown that mobile applications increase patient awareness, self-evaluation skills, and self-management abilities (Tang et al., 2020).

Mobile learning allows individuals to access information, interact with others, and receive instant feedback without time or location constraints (Bulut Özek & Gür, 2021). Mobile health interventions offer several advantages, including improved disease management, enhanced preventive care, effective monitoring of chronic conditions, reduced costs, and increased patient autonomy (Gruessner, 2015; Ardahan et al., 2018). Despite growing evidence supporting mobile health interventions, studies specifically examining the effect of mobile education on comfort levels in individuals living with a stoma remain limited. Therefore, this study aims to evaluate the effect of a comfort theory-based mobile education program on the comfort levels of individuals living with a stoma.

Type of the study: It is planned as a randomized controlled experimental and single-blind study.

Study setting(s): The study will be conducted in the urology and general surgery units of Izmir City Hospital.

Study Population / Sample

The population of the study will consist of patients who are hospitalized in the urology and general surgery units of Izmir City Hospital and are scheduled to undergo ostomy surgery between January 2026 and May 2026. The sample of the study will consist of patients who were hospitalized in the urology and general surgery units of Izmir City Hospital between January 2026 and May 2026, who meet the sample selection criteria of the study and who agree to participate in the research.

Considering the sample selection criteria, the study will include two groups, an experimental group and a control group. In order to determine the sample size, a power analysis was conducted using the G*Power 3.1.7.9 program to evaluate the comfort levels of ostomy patients and to determine the effect of education provided through a mobile education program based on Kolcaba's Comfort Theory on comfort levels. Since no similar reference study could be identified, the effect size determined by Cohen was used for the power analysis. Based on the power analysis calculated according to the difference between the experimental and control groups, with an alpha value of 0.05, an effect size of 0.8, and a theoretical power of 90%, the minimum sample size was calculated as 68 participants (34 in the experimental group and 34 in the control group). Patients will be assigned to the study groups using a computer-based randomization program (https://www.random.org/).

Hypothesis(es):

H0: Mobile education based on Kolcaba's Comfort Theory does not affect the comfort levels of patients with a stoma.

H1: Mobile education based on Kolcaba's Comfort Theory affects the comfort levels of patients with a stoma.

Data Collection Method

In data collection, the Patient Identification Form, the General Comfort Questionnaire, and a mobile education program including an animation video explaining stoma care for patients with a stoma based on Kolcaba's Comfort Theory will be used.

General Comfort Questionnaire

The General Comfort Questionnaire was developed by Kolcaba in 1992. The Turkish validity and reliability study was conducted by Kuğuoğlu and Karabacak in 2008. The scale consists of 48 items and three subdimensions (relief, ease, and transcendence) and is scored using a four-point Likert scale. The questionnaire includes both positively and negatively worded items, with negative items being reverse-coded during analysis.

The total score obtained from the scale is divided by the number of items to calculate the mean score. The minimum possible score is 48 and the maximum possible score is 192. According to the mean comfort scores, 0-48 indicates poor comfort, 49-96 indicates moderate comfort, 97-144 indicates good comfort, and 145-192 indicates very good comfort. Higher scores indicate higher levels of comfort. The Cronbach's alpha coefficient of the Turkish version of the scale is 0.85 (Kolcaba, 2003; Kuğuoğlu & Karabacak, 2008).

Mobile Education Content for Patients With a Stoma Based on Kolcaba's Comfort Theory and Development Stages

The design process of the mobile application developed for patients with a stoma will be planned in five stages. These stages include Analysis, Design, Development, Implementation, and Evaluation.

Stage 1: Analysis Phase of the Mobile Application

This is the initial stage in which the purpose of the mobile application is determined. The mobile application development process begins with the analysis phase, during which the goals and scope of the project are defined. Based on a comprehensive literature review focusing on factors affecting adaptation to life with a stoma, improvement of quality of life, and enhancement of comfort levels, the content of the mobile application will be developed.

The cost and software requirements of the mobile application will also be determined during this phase. Costs will include content development, animation-based video production, and mobile application software development. Content costs may vary depending on the use of photographs, videos, animations, and other materials. The application content will be supported by an animation-based nursing stoma care education video.

The mobile application will not include any diagnostic or treatment methods; it will only contain an animation-based nursing stoma care education video developed for patients with a stoma. The application will operate on both Android and iOS platforms to reach a wider user population. The software development process will focus on a simple menu structure and easily accessible content. Software costs will depend on database complexity, language support, mobile license requirements, and the scope of in-app functions. User data security, protection of personal information, and system performance sustainability will also be analyzed during this phase.

At the end of the analysis phase, a preliminary prototype of the mobile application will be developed based on content and functional requirements and submitted for expert review.

Stage 2: Design Phase of the Mobile Application

During the design phase, the basic visual and functional components of the application, including content layout, user interface, and user experience, will be structured. Collaboration will be established with professionals specialized in graphic design and software development to create a professional infrastructure.

A graphic designer will be consulted for the creation of the application logo. A computer programmer and a computer engineer will collaborate to transfer content related to stoma definition, types of stomas, risk factors, postoperative nursing care, and complication prevention into the mobile application. The application will include the following main sections: logo, login screen, registration screen, home screen, care video screen, care reminder screen, basic stoma information screen, contact screen, about us screen, and evaluation screen.

Stage 3: Mobile Application Development Phase

The application content will be developed based on guidelines published by the Wound, Ostomy and Continence Nurses Society (WOCN), World Council of Enterostomal Therapists (WCET), European Association of Urology Nurses (EAUN), Turkish Ostomy Surgery Association, and the Stoma, Wound, Ostomy and Incontinence Nurses Association, as well as relevant literature.

Mobile education content will be prepared in accordance with Kolcaba's Comfort Theory. The animation-based educational video will be developed using this theoretical framework. The main topics covered in the educational video include stoma definition, postoperative stoma care, stoma complications, indications for emergency department referral, symptom management, and comfort-enhancing care strategies.

The animation-based educational video will visually model nursing practices and allow patients to follow the care process step by step. Based on Kolcaba's Comfort Theory, the physical, psychospiritual, environmental, and sociocultural comfort needs of individuals with a stoma will be analyzed, and relevant educational content will be integrated into the application modules. No diagnostic or treatment methods will be included in the mobile application.

Stage 4: Implementation and Usability Testing of the Mobile Application 4.1 Pilot Testing

A pilot test will be conducted with three individuals with a stoma prior to field implementation. These individuals will not be included in the study sample and will only be involved in evaluating technical functionality, content accessibility, and user experience. During the pilot phase, the following aspects will be assessed:

Application launch speed, page transitions, and video playback functionality

Comprehensibility of educational content

Identification and revision of technical issues and usability challenges based on feedback

4.2 Inclusion of Participants in the Application

After obtaining informed consent, the mobile application will be installed on the smartphones of participants included in the study sample.

Individual face-to-face training on application use will be provided by the researcher

Core functions such as home screen navigation, module access, video viewing, and care reminder usage will be explained

Participants will be free to use the application at their own pace and frequency

4.3 Usage Process and Monitoring

Participants will be encouraged to actively use the mobile application throughout the specified study period. During this time:

In-app progress (completed modules) will be monitored through built-in analytics

The researcher will periodically contact participants to record feedback, problems, or suggestions

4.4 Ethical Principles and Data Security

Personal data will not be collected through the application; only content usage will be monitored

All information related to application usage will be kept confidential and not shared with third parties

Participants may withdraw from the study at any time

The usability of the mobile application will be evaluated using the Mobile Application Usability Scale (Appendix III). The Turkish validity and reliability study of this scale was conducted by Güler (2019). The scale consists of 40 items across 10 factors, each containing four items, and uses a seven-point Likert scale.

To evaluate the reliability and information quality of the animation-based educational content, an expert opinion form developed by the researcher will be used.

Randomization and Intervention Process

Participants will be assigned to experimental and control groups using a simple randomization method. Randomization will be performed using computer-generated random numbers, ensuring equal probability of group assignment for each participant (https://www.random.org/

).

Experimental Group

After explaining the purpose of the study, written informed consent will be obtained from participants assigned to the intervention group. The initial meeting will be conducted within the first 24 hours after hospital admission. One day before surgery, the Patient Identification Form and the General Comfort Questionnaire will be administered as pretests.

After baseline assessment, the mobile education program based on Kolcaba's Comfort Theory will be delivered individually in a single session lasting no longer than 30-45 minutes in a quiet hospital room. The control group will receive standard care.

On postoperative day one, both groups will be reassessed using the General Comfort Questionnaire. The intervention group will receive the mobile education again, while the control group will continue with standard care.

Fifteen days after hospitalization, participants will be contacted by phone to answer questions related to the educational content, and the General Comfort Questionnaire will be administered again (10-15 minutes). One month after hospitalization, a final face-to-face assessment will be conducted during the outpatient clinic visit, after which patient follow-up will be concluded (Wang et al., 2019; Vicdan, 2020).

Control Group

Written informed consent will be obtained from participants assigned to the control group. The initial meeting will occur within the first 24 hours after hospital admission. One day before surgery, the Patient Identification Form and the General Comfort Questionnaire will be administered as pretests.

No additional education will be provided to the control group by the researcher. Participants will receive routine hospital care during hospitalization. Comfort levels will be reassessed on postoperative day one, day fifteen via phone call, and at one month during the outpatient clinic visit. After completion of final data collection, the mobile education program based on Kolcaba's Comfort Theory will also be provided to the control group.

Statistical Analysis

Data collected in accordance with the study objectives will be analyzed using the Statistical Package for the Social Sciences (SPSS) version 22.0. Descriptive statistics will be presented as mean, standard deviation, minimum-maximum values, and percentages. Data normality will be assessed using the Kolmogorov-Smirnov and Shapiro-Wilk tests.

For normally distributed data, the independent samples t-test will be used to compare two groups. For non-normally distributed data, the Mann-Whitney U test will be used for two-group comparisons, and the Kruskal-Wallis test will be applied for comparisons involving three or more groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Patients with a stoma (colostomy or urostomy)
* Ability to use a smartphone or mobile device
* Willingness to participate in the study
* Ability to provide informed consent

Exclusion Criteria:

* Cognitive impairment that prevents understanding of the study procedures
* Severe psychiatric disorders
* Inability to use mobile technology
* Participation in another interventional study during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comfort Level of Patients with a Stoma | Preoperative period, postoperative day 1, postoperative day 15, and 1 month after surgery
  The comfort level of patients with a stoma will be measured using the General Comfort Questionnaire developed by Kolcaba. The scale assesses overall comfort across physical, psychospiritual, sociocultural, and environmental dimensions. Total comfort scores will be compared between the intervention and control groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Liao W, Chen X. Effects of a Short-term Mindfulness-Based Intervention on Comfort of Stroke Survivors Undergoing Inpatient Rehabilitation. Rehabil Nurs. 2019 Mar/Apr;44(2):78-86. doi: 10.1097/rnj.0000000000000098. PMID 30830883
- [Background] Hsu, M. Y., et al. (2020). Preoperative stoma site marking decreased stoma and peristomal complications. Journal of Wound Ostomy & Continence Nursing. https://doi.org/10.1097/WON.0000000000000634 Kang, Y., et al. (2025). Life experience of patients living with urostomy: A meta-synthesis. Psycho-Oncology, 34, e70096. https://doi.org/10.1002/pon.70096 Karadağ, A., et al. (2011). Ostomili bireylere yönelik uyum ölçeğinin Türkçeye uyarlanması. Ulusal Cerrahi Dergisi, 27(4), 206-211. Kolcaba, K. (1992). Holistic comfort: Operationalizing the construct as a nurse-sensitive outcome. Advances in Nursing Science, 15(1), 1-10. Kolcaba, K. (2003). Comfort theory and practice: A vision for holistic health care and research. Springer. Kuğuoğlu, S., Karabacak, Ü. (2008). Genel konfor ölçeğinin Türkçe'ye uyarlanması. İ.Ü.F.N. Hemşirelik Dergisi, 16(61), 16-23. Kuzu, M. A., et al. (2002). Effect of sphincter-sacrificing surgery for rectal carcinoma on quality of life. Diseases of the Colon & Rectum, 45(10), 1359-1366. Langer, A., et al. (2021). Digital health and remote interventions. NPJ Parkinson's Disease, 7(1). https://doi.org/10.1038/S41531-021-00160-3 Pinquart, M., Duberstein, P. R. (2010). Depression and cancer mortality: A meta-analysis. Psychological Medicine, 40(11), 1797-1810. Salvadalena, G. (2013). The incidence of stoma and peristomal complications. Journal of Wound, Ostomy and Continence Nursing, 40(4), 400-406. https://doi.org/10.1097/WON.0b013e318295a12b
- [Background] Barnwell, A. (2015). Advanced nursing practice in colorectal and stoma care. Gastrointestinal Nursing, 13(1), 42-48. https://doi.org/10.12968/gasn.2015.13.1.42 Brady, R. R. W., et al. (2025). The prevalence of leakage, peristomal skin complications and impact on quality of life in the first year following stoma surgery. Nursing Reports, 15, 107. https://doi.org/10.3390/nursrep15030107 Bulut Özek, M., Gür, D. (2021). Mobil öğrenmenin öğrencilerin akademik başarısı, motivasyonu ve tutumları üzerine etkisi: Bir meta-analiz. Trakya Eğitim Dergisi, 11(1), 1-15. https://doi.org/10.24315/tred.581539 Burch, J. (2015). Examining stoma care guidance for nurses. Gastrointestinal Nursing, 13(6), 17-25. https://doi.org/10.12968/gasn.2015.13.6.17 Çınar Yücel, Ş. (2011). Kolcaba'nın konfor kuramı. Ege Üniversitesi Hemşirelik Yüksekokulu Dergisi, 27(2), 79-88. Duluklu, B., Çelik, S. Ş. (2019). Kolostomisi olan bireylerde yaşam kalitesi: Sorunlar ve hemşirelik girişimleri. HUHEMFAD-JOHUFON, 6(2), 111-119. Goldberg, M., et al. (2018). WOCN Society clinical guideline: Management of the adult patient with a fecal or urinary ostomy. Journal of Wound, Ostomy and Continence Nursing, 45(1), 50-58. https://doi.org/10.1097/WON.0000000000000396 Grant, M., et al. (2013). Development of a chronic care ostomy self-management program. Journal of Cancer Education, 28, 70-78. Gruessner, V. (2015). The advantages of mobile health apps today and tomorrow. https://mhealthintelligence.com
- [Background] Akalın, B., Modanlıoğlu, A. (2020). 'Ameliyathane hemşiresi olmak': Nitel bir çalışma. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 23(1), 100-108. Aksoy, G., Çavdar, İ. (2015). Sindirim sistemi (gastrointestinal sistem) stomalarında bakım. In N. Akyolcu & N. Kanan (Eds.), Yara ve Stoma Bakımı (1. Baskı, ss. 67-81). Nobel Tıp Kitapevleri. Aminisani, N., Nikbakht, H., Jafarabadi, M. A., & Shamshirgaran, S. M. (2017). Depression, anxiety, and health-related quality of life among colorectal cancer survivors. Journal of Gastrointestinal Oncology, 8(1), 81-88. https://doi.org/10.21037/jgo.2017.01.12 Ayalon, R., Bachner, Y. G. (2019). Medical, social, and personal factors as correlates of quality of life among older cancer patients with permanent stoma. European Journal of Oncology Nursing, 38, 50-56. https://doi.org/10.1016/j.ejon.2018.11.010 Ayaz, S. (2008). Stomalı bireylerin cinsel sorunlarına yaklaşım. Türkiye Klinikleri Journal of Medical Ethics, 16, 89-93. Ayık, C., Özden, D. (2023). Stoma komplikasyonları ve hemşirelik bakımı: Güncel yaklaşımlar. Etkili Hemşirelik Dergisi, 16(3). Ayık, C., Özden, D., Cenan, D. (2020). Ostomy complications, risk factors, and applied nursing care. Wound Management & Prevention, 66(9), 20-30. https://doi.org/10.25270/wmp.2020.9.2030